CLINICAL TRIAL: NCT06605274
Title: Web-based Training Given to Women Who Have Experienced Perinatal Loss the Effect of Psychosocial Well-being
Brief Title: Effectiveness Web-based Training on Perinatal Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Nevin Çıtak BİLGİN, Assoc. Prof, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AIBU-SBF-NB-01
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Pregnancy Loss; Psychological Distress; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Prospective parallel two group unmasked prevention study
Masking Description: no masking used in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-Based Education Group (Other): The technology-based education program prepared for women experiencing perinatal loss was prepared based on current literature and care theories related to perinatal loss. The program consisted of five modules, namely "What I am experiencing, I am ready to learn", "I have a loss and I am ready to experience my mourning process", "I am experiencing my loss and I do not have to be alone", "I am ready to look back and explore", and "create a memory, move on". Expert opinions were obtained for the content of the program. Necessary adjustments were made to the program in line with expert opinions.
  Interventions: Other: Web-Based Education Program
- Control Group (Active Comparator): A conventional post discharge follow up was performed on control group no other intervention was applied.
  Interventions: Other: Control

INTERVENTIONS:
Other: Web-Based Education Program — Before being discharged from the clinic, the women who experienced perinatal loss filled out the Personal Information Form, Perinatal Grief Scale, Edinburgh Postnatal Depression Scale, Beck Hopelessness Scale, and Stress Coping Styles Scale individually. The women were informed about the use of the website. The discharged women were contacted by phone, given the passwords of the "birliktegücleniyoruz.com" website, and invited to use the website for the five-week education program. Each week, only one session determined for that week was uploaded to the site. Participants who wished to do so were able to watch the uploaded sessions more than once. Retrospective sessions also remained accessible on the site. Each session lasted an average of 20-30 minutes. Women who completed five sessions were contacted by phone in the sixth week. Women filled out the PGS, EPDS, BHS, and SCSS online a second time
  Arms: Web-Based Education Group
Other: Control — Before being discharged from the perinatology clinic, the women filled out the Personal Information Form, PGS, EPDS, BHS, and SCSS individually. Six weeks after discharge, the participants filled out the same measurement tools online again. During this process, the hospital's routine monitoring continued for the control group. The website was opened to the use of participants who wanted to use the site after the completion of the final tests.
  Arms: Control Group

SUMMARY:
The study was conducted in a randomized controlled parallel group experimental design to determine the effect of web-based supportive care provided to women who experienced perinatal loss on perinatal grief, depression, hopelessness and coping with stress.

DETAILED DESCRIPTION:
Loss, which includes many complex emotions, is the loss of a person or object that is valuable to the individual after having it. Perinatal loss is the most painful situation that pregnancy can potentially result in. With perinatal loss, parents may show behavioral (shock, anger and loneliness) and physical (crying, loss of appetite or overeating, insomnia, irritability, inability to concentrate, forgetfulness, pain, etc.) reactions. However, emotional problems such as grief and depression after loss are more common than physical and behavioral problems. While the prevalence of major depression in society is 3-10%, this rate varies between 10-51% in those who experience perinatal loss. Loss can become a life crisis with biopsychosocial and spiritual dimensions for parents and especially for women.

ELIGIBILITY:
Inclusion Criteria:

* spoke Turkish, had at least primary school level education
* did not have a psychiatric disease diagnosis
* could use and access the internet and information technologies
* did not have vision and hearing problems
* experienced pregnancy loss of 12 weeks or more
* were hospitalized in the perinatology clinic

Exclusion Criteria:

* Women who did not accept to participate in the study
* did not use the internet and information technologies and could not access them
* applied to psychological support units during the training process
* started using psychiatric medication during the training process were not included in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Perinatal Grief Scale (PGS) | six weeks
  The scale that evaluates the grief experienced after perinatal loss was developed by Toedter et al. The validity and reliability of the Turkish version of the scale was performed by Köneş et al. PGS consists of three sub-dimensions and is a 5-point Likert type.
Edinburgh Postnatal Depression Scale (EPDS) | six weeks
  The scale was developed by Cox and Hodden to determine the risk of postnatal depression. Its Turkish adaptation was made by Engindeniz et al. EPDS consists of 10 items and is a 4-point Likert type. The items are scored between 0-3.
Beck Hopelessness Scale (BHS) | six weeks
  It was developed by Beck, Trexler and Lester to determine individuals' hopelessness about the future. Its Turkish validity and reliability study was conducted by Seber et al. The scale consists of 20 items and three sub-dimensions. Scale items are scored between 0-1.
Stress Coping Styles Scale (SCSS) | six weeks
  The scale was created by Folkman and Lazarus to determine individuals' coping with stress. It was adapted to Turkish by Şahin and Durak. The scale consists of 30 items, five sub-dimensions, and is a 4-point Likert-type scale. The items in the scale are scored between 0 and 3. The sub-dimensions of the scale are "self-confident approach", "optimistic approach", "submissive approach", "helpless approach" and "seeking social support". The score obtained from the relevant sub-dimensions indicates that the individual uses the mentioned approach more

CONTACTS AND LOCATIONS:
Overall Officials: Nevin Bilgin, PhD, Study Director — Abant Izzet Baysal University; Tuba Ünal, Msc, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no data sharing plan was determined